CLINICAL TRIAL: NCT05283187
Title: The Effect of Mindfulness-Based Cognitive Therapy Program (MBCT) Applied to Nursing Students on Depression, Anxiety, Stress and Cognitive Flexibility: A Randomized Controlled Study
Brief Title: The Effect of Mindfulness-Based Cognitive Therapy Program Applied to Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Ferhan Acikgoz, Lecturer, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DuzceUFAcikgoz1
Record Dates: First submitted 2021-12-13; First posted 2022-03-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Mindfulness; Depression, Anxiety; Stress; Nursing Students
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT (Experimental): Mindfulness Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy Group
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy Group — Mindfulness Based Cognitive Therapy
  Arms: MBCT

SUMMARY:
Among the stress factors of nursing students are traumatic experiences such as death and encountering a dying patient from the first moments of their education years, fear of making mistakes in the clinic, patient care, not getting enough support from the instructor or clinic staff, and communication problems. Exposure to long-term and uncontrollable stress negatively affects students' professional identity development and health. Students who cannot cope with their stress feel stress at a higher level and as a result they may experience anxiety and depression.It is important for nurse candidates to graduate by being supported in all aspects, both in terms of individual and professional development. For this reason, nursing educators should use effective and innovative interventions to help students recognize the stress they experience and help them reduce stress. Mindfulness-Based Cognitive Therapy Program (MBCT) is one of these programs. Although studies with MBCT are found in the literature, our country In the literature, no randomized controlled studies were found with nursing students. In line with this information, it was thought that mindfulness-based studies were needed. This study was planned to determine the effect of MBCT program on depression, anxiety, stress and cognitive flexibility of nursing students.

DETAILED DESCRIPTION:
Inclusion criteria for research

* to be nursing students
* to have a score of 4 or more (General Health Questionnaire)
* Internet access to participate in online sessions
* Individuals who voluntarily agree to participate in the research will be included.

Exclusion criteria from the research

* Those who are in the acute depression period
* Risk of suicidal
* Having participated in MBSR-MBCT programs before

Application Protocol Principles

* to consider students individuality, to provide correct information/education,
* Guiding to increase motivation,
* Giving feedback and supporting individuals,
* to provide accessibility for individuals' concerns and questions,

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Düzce University, Faculty of Health Sciences, Department of Nursing
* Individuals who voluntarily agree to participate in the research

Exclusion Criteria:

* Those in acute depression

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Depression at 3 Months | Baseline and 8 week and 12 week
  Depression Stress and Anxiety Scala-42 (depression score; first to nine normal, 10-13 mild, 14-20 is intermediate, 21-27 is advanced, over 28 is very advanced)

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Karaca, Study Director — Duzce University; Ferhan Açıkgöz, Principal Investigator — Duzce University
Locations (1):
- Ferhan Açıkgöz, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuksel A, Bahadir-Yilmaz E. Relationship between depression, anxiety, cognitive distortions, and psychological well-being among nursing students. Perspect Psychiatr Care. 2019 Oct;55(4):690-696. doi: 10.1111/ppc.12404. Epub 2019 May 29. PMID 31140627